CLINICAL TRIAL: NCT05916430
Title: Community-viable Screening for Autism Spectrum Disorder (ASD) in 9-month-old Infants Using Quantitative Eye-tracking Assays of Social Visual Engagement
Brief Title: Screening for Autism in 9-Month-Olds by Measuring Social Visual Engagement
Status: Recruiting | Type: Observational
Sponsor: Emory University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Warren R. Jones, Associate Professor, Emory University
Other Study IDs: IRB00115022; 5R01MH121363-03 (NIH)
Record Dates: First submitted 2023-06-14; First posted 2023-06-23 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Autism; Infant Development
Keywords: Screening; well-baby visits; Social Development; Communicative Development; Development Disabilities; Autism Spectrum Disorders
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder | interventions — Early Detection of Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- General Population Screening Cohort: A general population cohort of 9-month-old infants presenting for well-child visits will be screened initially at 9 months of age, and then screened again sequentially at 12, 15, 18, 21, and 24 months, to test screening performance relative to outcome status with autism or developmental disabilities.
  Interventions: Diagnostic Test: EarliPoint Investigational Device

INTERVENTIONS:
Diagnostic Test: EarliPoint Investigational Device — Infants will complete eye-tracking data collection at the age of 9 months on the EarliPoint Investigational Device. Eye-tracking video cameras will safely measure the movements of the child's eyes while they watch age-appropriate video scenes of other children playing together. Parents/Caregivers will complete screening forms and questionnaires about their baby's health and development. Parents/caregivers will complete surveys about their child's development. The surveys will be emailed, to be completed when the child is approximately 9, 12, 15, 18, 21, and 24 months old. If the child shows signs of developmental delay, the child will be asked to participate in a comprehensive developmental and diagnostic assessment.
  Other Names: Screening test

SUMMARY:
The goal of this project is to measure the clinical utility of an objective and quantitative eye-tracking assay collected on a standalone, mobile investigational device to accurately screen 9-month-old infants for autism spectrum disorder and other actionable delays.

DETAILED DESCRIPTION:
The purpose of this study is to see if measuring how infants look at social information can be used as a screening tool to identify developmental delays or vulnerabilities in infants as young as 9 months of age. What the 9-month-old infant looks at will be measured with eye-tracking technology, which uses a video camera to safely measure the child's eye movements while the child watches video scenes of other children at play. Parents/caregivers will be asked if they would like to participate during their child's 9-month well-baby visit at their pediatrician's office. If they agree to participate, the child will have their first study visit at this time. Children will undergo an eye-tracking session to measure social looking. Parents/caregivers will also complete forms and questionnaires about their child's health and development. The forms will be emailed, to be completed when the child is approximately 9, 12, 15, 18, 21, and 24 months old.

If a child shows signs of developmental delay (DD) or autism spectrum disorder (ASD), the child will be asked to participate in a comprehensive developmental and diagnostic assessment in-person with expert clinicians when the child is between 18-26 months old, to determine the child's strengths and any vulnerabilities, and to recommend any support or treatment if needed.

If the child does not show signs of developmental delay and/or autism, the investigators may still invite the child for an in-person assessment with expert clinicians when the child is between 18-26 months old. Approximately 10% of children who do not show any signs of developmental delay and/or autism will be randomly selected for an in-person assessment. At the end of the assessment, parents/caregivers will be provided feedback on their child's strengths and any vulnerabilities and, if necessary, a report will be written to help them access services for their child.

ELIGIBILITY:
Inclusion Criteria:

* Infants between the chronological ages of 8-10 months
* Infants must be generally healthy with no acute illnesses likely to prevent successful or valid data collection (e.g., current vomiting, high fever, conjunctivitis affecting vision)
* Participants' parents/caregivers must be able to understand and voluntarily provide written informed consent.

Exclusion Criteria:

- Children will be excluded if they have signs of acute illness likely to prevent successful or valid data collection (e.g., conjunctivitis affecting vision, current vomiting, or high fever).

Ages: 8 Months to 10 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants presenting for a 9-month well-child visit between the chronological ages of 8-10 months with no acute illnesses
Sampling Method: Probability Sample
Enrollment: 2120 (Estimated)
Dates: Start 2023-02-02 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Accuracy of eye-tracking assays at 9 months relative to ASD vs. non-ASD diagnosis at 24 months | 24 months
  Diagnostic performance measured by sensitivity, specificity, area under the receiver operating characteristic curve, positive predictive value, and negative predictive value of the eye-tracking-based assays when compared with clinical reference standard diagnostic outcome of ASD or non-ASD.
Accuracy of eye-tracking assays at 9 months relative to Affected (ASD or DD) vs. Unaffected status at 24 months. | 24 months
  Diagnostic performance measured by sensitivity, specificity, area under the receiver operating characteristic curve, positive predictive value, and negative predictive value of the eye-tracking-based assays when compared with clinical reference standard diagnostic outcome of Affected vs. Unaffected.

SECONDARY OUTCOMES:
Measure the ability of eye-tracking assays at 9 months to predict dimensional levels of social disability at 18-26 months compared to the Autism Diagnostic Observation Schedule, 2nd Edition (ADOS-2) | 18-26 months
  Eye-tracking assays at 9 months will generate a social disability index; investigators will measure the correlation between that index and results on a standardized assessment by the ADOS-2 of autistic social disability conducted by expert clinicians at 18-26 months.
Measure the ability of eye-tracking assays at 9 months to predict dimensional levels of verbal ability at 18-26 months compared to the Mullen Scales of Early Learning | 18-26 months
  Eye-tracking assays at 9 months will generate verbal ability indices; investigators will measure the correlation between those indices and results from a standardized assessment of expressive and receptive language function (the Mullen Scales of Early Learning). Receptive Language and Expressive Language Scales of the Mullen Scales of Early Learning (standardized measures of language function). Each item within these scales is scored either from 0 to 5 points for certain items or as 0 (skill not demonstrated) or 1 (correct response) for others. Raw scores are calculated by summing item-level ratings from the basal to the ceiling item. These raw scores are converted to standardized T-scores for analysis and interpretation (range: approximately 20-80 T-score; mean = 50, SD = 10; higher scores = better performance). The MSEL also yields an Early Learning Composite (mean = 100, SD = 15; higher scores = better overall performance).
Measure the ability of eye-tracking assays at 9 months to predict dimensional levels of nonverbal cognitive ability at 18-26 months. | 18-26 months
  Eye-tracking assays at 9 months will generate nonverbal ability indices. Investigators will assess the correlation between those indices and results from the Visual Reception Scale of the Mullen Scales of Early Learning (a standardized measure of nonverbal cognitive function). Each item on the Visual Reception Scale is scored either from 0 to 5 points for certain items or as 0 (skill not demonstrated) or 1 (correct response) for others. Raw scores are calculated by summing item-level ratings from the basal to the ceiling item. These raw scores are converted to standardized T-scores for analysis and interpretation (range: approximately 20-80 T-score; mean = 50, SD = 10; higher scores = better performance).

CONTACTS AND LOCATIONS:
Overall Officials: Warren R Jones, PhD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Emory University, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Yes
Data are planned to be publicly reposited in the NIMH Data Archive (https://nda.nih.gov) after publication, with accession number added when available.
Time Frame: After publication
Access Criteria: Access will follow standard NIMH NDA processes, as detailed on the website: https://nda.nih.gov/nda/faq.html